CLINICAL TRIAL: NCT03593057
Title: Effectiveness of a Manual Therapy Protocol in Women With Dysmenorrhea
Brief Title: Effectiveness of Manual Therapy in Dysmenorrhea
Acronym: MTDysmen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, GEMMA V ESPÍ LÓPEZ, PhD, Principal Investigator, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ID0023
Record Dates: First submitted 2018-06-01; First posted 2018-07-19 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Dysmenorrhea Primary
Keywords: dysmenorrhoea; manual therapy
MeSH Terms: conditions — Dysmenorrhea | interventions — Musculoskeletal Manipulations; Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual therapy protocol (Experimental): Manual therapy protocol and self-care advice and body awareness. Three sessions of manual therapy will be applied, (at the beginning, at 2 weeks and at 3 weeks).
  Interventions: Other: Control group
- Control group. (Active Comparator): Advice on self-care and body awareness.
  Interventions: Other: Manual therapy

INTERVENTIONS:
Other: Manual therapy — Manual therapy protocol and self-care advice and body awareness.
  Arms: Control group.
Other: Control group — Advice on self-care and body awareness.
  Arms: Manual therapy protocol

SUMMARY:
The objective of this clinical study would be to verify if manual therapy is effective in the treatment to reduce pain in women suffering from primary dysmenorrhea.

Material and methods In this experimental study, women diagnosed with primary dysmenorrhea will be included, which will be divided randomly into two groups: an intervention group and a comparator group.

The study will last nine weeks (3 menstrual cycles). Patients in the intervention group will receive 3 treatment sessions.

The evaluation will include pain, the quality of life, the global impression of change, personal body satisfaction and global self-perception and the pain perception.

DETAILED DESCRIPTION:
Introduction The prevalence of primary dysmenorrhoea is high and has an impact on quality of life, pain and disability. The cause is due to the increase of postaglandins that can be influenced by the lowering of progesterone. In short, there is a complex relationship between hormones and the immune system.

Manual therapy increases the mobility of the sacrum and tissues of the pelvis, increasing the blood supply and the uterus that has parasympathetic innervation through the sacrum improves mobility, motility and irrigation.

The ligaments, fasciae and tissue of the pelvis improve their irrigation through fascial, mobility and visceral techniques, which would improve uterine mobility by anatomical connections with these structures. With better mobility the uterus, and therefore the smooth muscle, would have more irrigation and less pain and hypercontractivility.

The adjacent tissues, perineum, triangular ligament, innervated by the vagus nerve, improve

The main objective is the improvement of quality of life, personal body satisfaction and overall self-perception and pain reduction in women with dysmenorrhea after treatment with manual therapy and provide information and advice on self-care and menstrual awareness.

Methods

Sample. The sample is formed by women with dysmenorrhoea aged between 18 and 45 years, with no other abdominopelvic problems.

Design. The sample will be divided into 2 groups: Group 1. Manual therapy protocol and self-care advice and body awareness. Three sessions of manual therapy will be applied, (one at the beginning, another at 2 weeks and another at 3 weeks); Group 2 comparator. Advice on self-care and body awareness.

Evaluations:

* Clinical interview with anthropometric data and characteristics of the pathology (age, weight, height, pain characteristics) There will be 3 evaluations: Evaluation at the beginning, at the end of the treatment and a follow-up of one month.
* SF-36 quality of life scale.
* Visual Analog Scale (EVA).
* Feeling of change after treatment with the Patient Global Impression of Change Scale.
* Personal Body Satisfaction and Global Self-Perception.
* McGill pain perception questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Women with menstrual pain of more than 6 months of evolution.
* Women with pain equal to or greater than 4 on the visual analogue scale in more than half of their one-year menstrual cycles.

Exclusion Criteria:

* Hormone treatment
* Contraindication to any of the treatments
* Participate in this period of no functional recovery program or physiotherapy treatment.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women with dysmenorrhoea
Enrollment: 39 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale of Pain. | 9 weeks
  The participants are asked to mark the intensity of pain from 1 to 10, with 1 being almost non-existent and 10 being the worst pain imaginable.

SECONDARY OUTCOMES:
SF-36 quality of life scale. | 9 weeks
  It consists of 36 items with the following scales: Physical function (items 3a, 3b, 3c, 3d, 3e, 3f, 3g, 3h, 3i, 3j), Physical role (items 4a, 4b, 4c, 4d), Corporal pain ( items 7, 8), General Health (items 1, 11a, 11b, 11c, 11d), Vitality (items 9a, 9e, 9g, 9i), Social function (items 6, 10), Emotional role (items 5a, 5b, 5c) and Mental Health (items 9b, 9c, 9d, 9f, 9h). Includes an item on the change in the general health status with respect to the previous year (item 2). To calculate the score, we must first homogenize the address of the answers by re-coding the items that require it, so that "the higher the score, the better the health condition", then the calculation of the sum of the items of each scale and, finally, the linear transformation of raw scores on a scale of 0 (worst health status for that dimension) to 100 (the best health status).
Global Impression Change Scale. | 9 weeks
  To assess the change perceived after the treatment, patients are asked to rate their perception of change in the Global Impression Change Scale of the patient, and a questionnaire with a question and 7 alternatives, being 1 "maximum change" and 7 "Nothing of change".
Body Satisfaction and global self-perception Questionnaire. | 9 weeks
  It contains 10 positive and 10 negative adjectives about the participant's body sensation with alternative answers ranging from 1 = Excellent to 5 = Poor. Each question is scored independently.
McGill pain perception questionnaire. | 9 weeks
  This questionnaire assesses quantitative and qualitative aspects of pain, such as location, quality, temporal properties and intensity.
  We use the short version, which consists of several clearly differentiated parts: Quality of pain that define the one with 66 words grouped into several categories that in turn form four large groups, pain assessment index (PRI): total and for each of the four areas (PRI), sensory, emotional PRI, valued PRI and miscellaneous PRI). The score is calculated adding that of each group of words that make up each category; b) Number of words chosen (NWC): sum of the number of pain characteristics selected by the patient; c) Pain intensity index (PPI): selected response of the item that explores this aspect.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Faculty of Physiotherapy, Valencia
  - Gemma V Espí López, Valencia